CLINICAL TRIAL: NCT05010785
Title: Ridge Splitting With Simultaneous Implant Placement Using i-PRF With Guided Bone Regeneration: a Randomized Clinical Trial
Brief Title: Ridge Splitting With Simultaneous Implant Placement Using i-PRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Dalia Rasheed Issa, principal investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-73
Record Dates: First submitted 2021-08-01; First posted 2021-08-18 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Ridge Splitting; i-PRF; Dental Implant
MeSH Terms: interventions — proliferation regulatory factors, human urine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- alveolar ridge splitting with GBR and i-PRF (Experimental): alveolar ridge splitting in combination with the use of GBR with i-PRF (sticky bone) with immediate implant placement
  Interventions: Procedure: Immediate implant placement and alveolar ridge splitting with GBR and i-PRF
- alveolar ridge splitting with GBR (Active Comparator): alveolar ridge splitting in combination with the use of GBR without i-PRF (sticky bone) with immediate implant placement
  Interventions: Procedure: Immediate implant placement and alveolar ridge splitting with GBR

INTERVENTIONS:
Procedure: Immediate implant placement and alveolar ridge splitting with GBR and i-PRF — Implant insertion and GBR for augmentation of the gap between buccal and lingual plate using bone graft mixed with i-PRF
  Arms: alveolar ridge splitting with GBR and i-PRF
Procedure: Immediate implant placement and alveolar ridge splitting with GBR — Implant insertion and GBR for augmentation of the gap between buccal and lingual plate
  Arms: alveolar ridge splitting with GBR

SUMMARY:
Sohn introduced the concept of sticky bone in which i-PRF is mixed with the granules of bone graft, leading to fabrication of growth factors-enriched bone graft matrix using autologous fibrin glue. This minimizes bone loss and accelerates tissue healing during healing period. The present study was conducted to evaluate the clinical and radiographic outcomes following the application of the alveolar ridge splitting in combination with the use of guided bone regeneration (GBR) with or without i-PRF (sticky bone), associated with immediate implant placement in patients with horizontally atrophic jaw bones.

ELIGIBILITY:
Inclusion Criteria:

* good general health at the time of surgery.
* at least 3 months of healing after tooth extraction.
* horizontally compromised alveolar ridges at least 10 mm high and 3 mm wide.

Exclusion Criteria:

* a vertical bone defect in the edentulous ridge.
* thick cortex in the labial/buccal with less cancellous bone inside
* obvious undercut on the labial/buccal side.
* uncontrolled periodontal conditions or other oral disorders.
* history of radiotherapy in the head and neck region.
* uncontrolled diabetes mellitus or other systematic disorders.
* smokers.
* Pregnancy.
* non-compliant patients.
* allergic reaction to the medications used

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Measurements of the amount of bone formation in millimeters around immediately placed dental implants | 9 months
  Measurements of the amount of bone formation in millimeters using GBR with or without the combined effect of i-PRF in the ridge splitting following immediate implant placement.

CONTACTS AND LOCATIONS:
Overall Officials: Dalia R Issa, PhD, Principal Investigator — Kafrelsheikh University
Locations (1):
- Faculty of Dentistry, Kafrelsheikh University, Kafr ash Shaykh, Egypt